CLINICAL TRIAL: NCT01310985
Title: A Pilot Trial of Pre-Operative Chemoradiotherapy Using Capecitabine (Xelodaâ), External Beam Radiation and Cetuximab (Erbitux®) Followed by Definitive Surgery in Patients With Localized (Non-Metastatic) Rectal Cancer
Brief Title: A Trial of Pre-Operative Chemoradiotherapy Using Capecitabine, Radiation & Cetuximab, in Rectal Cancer
Status: Completed | Type: Observational
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: RAC# 2071-051; RAC# 2071-051 (Other: KFSH&RC IRB)
Record Dates: First submitted 2011-03-06; First posted 2011-03-09 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2011-12

CONDITIONS: Colon Rectal Cancer Duke Stage Stageval
Keywords: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Cetuximab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Capecitabine (Xelodaâ), XRT & Cetuximab (Erbitux®) — Capecitabine (Xelodaâ), External Beam Radiation and Cetuximab (Erbitux®)
  Other Names: Capecitabine (Xelodaâ), XRT& Cetuximab (Erbitux®)

SUMMARY:
A Pilot Trial of Pre-Operative Chemoradiotherapy Using Capecitabine (Xelodaâ), External Beam Radiation and Cetuximab (Erbitux®) Followed by Definitive Surgery in Patients With Localized (Non-Metastatic) Rectal Cancer

DETAILED DESCRIPTION:
Its a pilot study of pre-op chemotherapy and RT utilizing CAPECITABINE, XRT and CETUXIMAB in pts with locally advanced rectal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Localized Non-Metastatic Rectal Cancer

Exclusion Criteria:

* Patients with diagnosis other than Localized Non-Metastatic Rectal Cancer

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Localized (Non-Metastatic) Rectal Cancer
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2008-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of pre-operative concurrent chemotherapy with capacitabine (Xeloda), weekly cetuximab (Erbitux), and external beam radiation. | For the duration of the experiment

SECONDARY OUTCOMES:
Evaluate efficacy of sphincter preserving surgery rate, local recurrence rate and the disease free and overall survival in patients. | For the duration of the experiment

CONTACTS AND LOCATIONS:
Overall Officials: Shouki Bazarbashi, M.D., Principal Investigator — KFSH & RC
Locations (1):
- Kfsh & Rc, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided